CLINICAL TRIAL: NCT03315845
Title: Neuraxial Anaesthesia: Does BMI Relate to Palpability of Bony Landmarks and Are Standard Needles a Suitable First Choice in Patients With BMI>30kg/m2
Brief Title: Neuraxial Anaesthesia: Does BMI Relate to Ease of Neuraxial Anaesthesia?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Maternity Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Moninne Creaney, Dr. Moninne Creaney, Specialist Registrar in Anaesthesia, National Maternity Hospital, Ireland
Other Study IDs: NationalMHI
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Neuraxial Ultrasound; Obstetric Anaesthesia
Keywords: BMI; obstetric anaesthesia; neuraxial anaesthesia; neuraxial ultrasound; difficult neuraxial anaesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Palpation of bony landmarks for neuraxial anaesthesia. — Manual palpation of anterior and posterior iliac crests; lumbar spinous processes; scapulae; and sacral cornua.
  Ultrasound of neuraxial anatomy to assess depth to epidural space.
  Other Names: Neuraxial ultrasound

SUMMARY:
Neuraxial anaesthesia can be more difficult and associated with more complications if the patient's bony landmarks are difficult to palpate. They are more likely to be difficult to palpate if a patient has a high Body Mass Index (BMI), (>30kg/m2). The depth that the spinal or epidural needle must be inserted is usually longer in these patients with high BMIs. We wish to palpate the backs of at least 100 such patients to see how many of them have impalpable bony landmarks. We then wish to use ultrasound to measure the distance from skin to the posterior epidural complex to discover if this length is longer than the standard needle length. If it is longer in the majority of people we study, we will recommend changing standard practice to start using a longer needle for all first attempts at neuraxial anaesthesia in this patient population.

DETAILED DESCRIPTION:
Complications rates including failure are higher in obese patients undergoing anaesthesia procedures. Anaesthetists have adopted the use of ultrasound to assist in overcoming these difficulties. Neuraxial ultrasound is proving to be beneficial in those patients in whom identification of interspinous spaces is difficult and most of these patients are obese.

In our institution, there is a 'standard practice' for neuraxial procedures, with a 'standard' needle used for first attempts (Whitacre 25G 90mm for spinal, Tuohy 18G 80mm for epidural). If the operator has not reached the desired space (spinal or epidural) with the needle inserted to 8cm, a longer needle is then considered for further attempts. This exposes the patient to at least one extra neuraxial needle insertion. Studies have shown that increased needle insertions and redirections are associated with increased complications.

We hypothesised that a large number of patients with BMI>30kg/m2 would have a depth of spinal/epidural space that is greater than the length of the 'standard' needle used. Therefore we suggest that practice should change to use the longer needle or a combined spinal-epidural on the first attempt in these patients.

To test our hypothesis, we will assess the ease of palpation of the following anatomical landmarks: anterior and posterior iliac crests; lumbar spinous processes; scapulae; and sacral cornua. We will then perform neuraxial sonography of the lumbar spine, measuring depth to epidural space. Finally we will measure waist circumference in those patients with BMI <30kg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Recorded BMI >30kg/m2; ability to give consent; non-emergency cases.

Exclusion Criteria:

* Previous metal work to lumbar spine.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Obstetric patients.
Study Population: Obstetric patients with BMI >30kg/m2, presenting in a non-emergency situation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-23 (Estimated); Primary Completion 2018-01-09 (Estimated); Study Completion 2018-01-09 (Estimated)

PRIMARY OUTCOMES:
Palpability of bony landmarks for neuraxial anaesthesia | 4 months
  The percentage of patients with BMI>30kg/m2 who have difficult or impalpable bony landmarks including: lumbar spinous processes; anterior and posterior iliac spines; scapulae; and sacral cornua.

SECONDARY OUTCOMES:
Ultrasonographic distance from skin to posterior epidural complex | 4 months
  To use sonography to measure the distance from skin to the dural complex in these patients and quantify the percentage whose distance is greater than the length of the standard needle.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin McKeating, Study Director — National Maternity Hospital, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arzola C, Mikhael R, Margarido C, Carvalho JC. Spinal ultrasound versus palpation for epidural catheter insertion in labour: A randomised controlled trial. Eur J Anaesthesiol. 2015 Jul;32(7):499-505. doi: 10.1097/EJA.0000000000000119. PMID 25036283
- [Background] Ansari T, Yousef A, El Gamassy A, Fayez M. Ultrasound-guided spinal anaesthesia in obstetrics: is there an advantage over the landmark technique in patients with easily palpable spines? Int J Obstet Anesth. 2014 Aug;23(3):213-6. doi: 10.1016/j.ijoa.2014.03.001. Epub 2014 Mar 12. PMID 24768303
- [Background] Srinivasan KK, Lee PJ, Iohom G. Ultrasound for neuraxial blockade. Med Ultrason. 2014 Dec;16(4):356-63. PMID 25463890
- [Background] Grau T, Leipold RW, Delorme S, Martin E, Motsch J. Ultrasound imaging of the thoracic epidural space. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):200-6. doi: 10.1053/rapm.2002.29239. PMID 11915069
- [Background] Carnie J, Boden J, Gao Smith F. Prediction by computerised tomography of distance from skin to epidural space during thoracic epidural insertion. Anaesthesia. 2002 Jul;57(7):701-4. doi: 10.1046/j.1365-2044.2002.02572_4.x. PMID 12059829
- [Background] Gnaho A, Nguyen V, Villevielle T, Frota M, Marret E, Gentili ME. Assessing the depth of the subarachnoid space by ultrasound. Rev Bras Anestesiol. 2012 Jul;62(4):520-30. doi: 10.1016/S0034-7094(12)70150-2. PMID 22793967
- [Background] Seligman KM, Weiniger CF, Carvalho B. The Accuracy of a Handheld Ultrasound Device for Neuraxial Depth and Landmark Assessment: A Prospective Cohort Trial. Anesth Analg. 2018 Jun;126(6):1995-1998. doi: 10.1213/ANE.0000000000002407. PMID 28858898
- [Background] Balki M, Lee Y, Halpern S, Carvalho JC. Ultrasound imaging of the lumbar spine in the transverse plane: the correlation between estimated and actual depth to the epidural space in obese parturients. Anesth Analg. 2009 Jun;108(6):1876-81. doi: 10.1213/ane.0b013e3181a323f6. PMID 19448216